CLINICAL TRIAL: NCT04386083
Title: COVID-19 Outcomes: A Retrospective Study of Neurological Manifestations and Associated Symptoms (The Philippine CORONA Study)
Brief Title: Neurologic Manifestations of COVID-19
Acronym: CORONA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of the Philippines (Other)
Collaborators: Asian Hospital and Medical Center, Muntinlupa City, Philippines (Unknown); Baguio General Hospital and Medical Center, Baguio City, Philippines (Unknown); Cagayan Valley Medical Center, Tuguegarao City, Philippines (Unknown); Capitol Medical Center, Quezon City, Philippines (Unknown); Cardinal Santos Medical Center, San Juan City, Philippines (Unknown); Chong Hua Hospital, Cebu City, Philippines (Unknown); De La Salle University Medical Center (Other); East Avenue Medical Center, Philippines (Other Government); Jose B. Lingad Memorial Regional Hospital, San Fernando, Pampanga, Philippines (Unknown); Jose R. Reyes Memorial Medical Center (Other Government); Lung Center of the Philippines (Other); Manila Doctors Hospital, Philippines (Unknown); Manila Medical Center, Philippines (Unknown); Makati Medical Center (Other); New Era General Hospital, Philippines (Unknown); Quirino Memorial Medical Center, Philippines (Unknown); Ospital ng Makati, Philippines (Unknown); Dr. Pablo O. Torre Memorial Hospital, Bacolod City, Philippines (Unknown); Philippine Heart Center (Unknown); Research Institute for Tropical Medicine, Philippines (Other Government); San Juan De Dios Educational Foundation Inc. - Hospital, Philippines (Unknown); San Lazaro Hospital, Philippines (Unknown); Southern Isabela Medical Center, Philippines (Unknown); St. Luke's Medical Center, Philippines (Other); St Lukes Medical Center, Bonifacio Global City, Philippines (Unknown); Southern Philippines Medical Center (Other); The Medical City, Philippines (Other); University of the East Ramon Magsaysay Memorial Medical Center, Inc, Philippines (Unknown); University of Santo Tomas Hospital, Philippines (Other); Veterans Memorial Medical Center, Philippines (Unknown); Dr. Jose N. Rodriguez Memorial Hospital and Sanitarium (Other); Zamboanga City Medical Center, Zamboanga City (Unknown); Western Visayas Medical Center, Iloilo City (Unknown); Northern Mindanao Medical Center, Cagayan de Oro City (Unknown); Vicente Sotto Memorial Medical Center, Cebu City (Unknown); Perpetual Succor Hospital, Cebu City (Unknown)
Responsible Party: Principal Investigator, Adrian Espiritu, Principal Investigator, University of the Philippines
Other Study IDs: RGAO-2020-0348
Record Dates: First submitted 2020-05-04; First posted 2020-05-13 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Coronavirus Disease 2019
Keywords: COVID-19; neurological manifestations; outcomes; cohort study
MeSH Terms: conditions — COVID-19; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 patients with neurologic manifestations: Patients with confirmed COVID-19 disease who presented with neurological symptoms or new-onset neurological disorders/complications
- COVID-19 patients without neurologic manifestations: Patients with confirmed COVID-19 disease who did not present with neurological symptoms or new-onset neurological disorders/complications

SUMMARY:
This study will determine the neurological profile and predictors of outcomes in patients with COVID-19 disease in the Philippines. It will also evaluate if there is significant difference between COVID-19 patients with neurological manifestations compared to those COVID-19 patients without neurological manifestations in terms of various prespecified clinical outcomes. Furthermore, the likelihood of these outcomes in COVID-19 patients with neurological manifestations compared to those without neurological manifestation will be determined in this study.

DETAILED DESCRIPTION:
This quantitative, retrospective, cohort study will determine the following: 1) demographic, clinical and neurological profile of patients with COVID-19 disease in the Philippines; 2) the frequency of neurological symptoms and new-onset neurological disorders/complications in patients with COVID-19 disease; 3) the neurological manifestations that are significant predictors of mortality, respiratory failure, duration of ventilator dependence, intensive care unit (ICU) admission, length of ICU stay, and length of hospital stay; 4) if there is significant difference between COVID-19 patients with neurological manifestations compared to those COVID-19 patients without neurological manifestations in terms of mortality, respiratory failure, duration of ventilator dependence, ICU admission, length of ICU stay and length of hospital stay; and 5) the likelihood of mortality, respiratory failure and ICU admission in COVID-19 patients with neurological manifestations compared to those without neurological manifestations.

ELIGIBILITY:
Inclusion Criteria:

* Cases confirmed by testing approved patient samples (i.e. nasal swabs, sputum, bronchoalveolar lavage fluid) employing the real-time reverse transcriptase polymerase chain reaction (RT-PCR) from COVID-19 testing centers accredited by the DOH;
* adult patients at least 19 years of age;
* male or female;
* cases with clinical symptoms and signs attributable to COVID-19 disease (i.e. respiratory as well as non-respiratory clinical signs and symptoms), with or without the availability of ancillary tests (i.e. complete blood count, chest x-ray); cases with disposition (i.e. discharged or died) at the end of the study period.

Exclusion Criteria:

* Pediatric patients ≤18 years
* Cases with conditions of diseases caused by other organisms (i.e. bacteria, other viruses, fungi, etc.) or caused by other pathologies unrelated to COVID-19 disease (i.e., trauma).

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with confirmed COVID-19 disease
Sampling Method: Non-Probability Sample
Enrollment: 1342 (Estimated)
Dates: Start 2020-06-10 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Mortality (binary outcome) | from admission until occurrence of mortality, assessed up to 6 months
  Defined as patients with confirmed COVID-19 who died
Respiratory failure (binary outcome) | from admission until occurrence of respiratory failure, assessed up to 6 months
  Defined as the patient with confirmed COVID-19 who experienced clinical symptoms and signs of respiratory insufficiency. Clinically, this condition may manifest as tachypnea, abnormal blood gases (hypoxemia or hypercapnia), signs of increased work of breathing, and requires oxygen supplementation

SECONDARY OUTCOMES:
Duration of ventilator dependence (continuous outcome) | day of intubation to day of extubation, assessed up to 6 months
  Defined as the number of days from initiation of assisted ventilation to extubation
Intensive care unit (ICU) admission (binary outcome) | admission to ICU admission, assessed up to 6 months
  Defined as the patients with confirmed COVID-19 who are admitted to an ICU or ICU-comparable setting

OTHER OUTCOMES:
Length of ICU stay (continuous outcome) | ICU admission to ICU discharge, assessed up to 6 months
  Defined as the number of days admitted in the ICU or ICU-comparable setting
Length of hospital stay (continuous outcome) | admission to hospital discharge, assessed up to 6 months
  Defined as the number of days from admission to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Adrian I Espiritu, MD, Principal Investigator — University of the Philippines
Locations (1):
- Philippine General Hospital - University of the Philippines Manila, Manila, Philippines

IPD SHARING:
Plan to Share IPD: Yes
Researchers may be able to request data through an official letter addressed to the Steering Committee of the "The Philippine CORONA Study" e-mailed to coronastudyph@gmail.com.
Supporting Information: Study Protocol
Time Frame: Data will be stored for 5 years after completion of the study.
Access Criteria: Data may be requested through an official letter addressed to the Steering Committee of the "The Philippine CORONA Study" e-mailed to coronastudyph@gmail.com.

REFERENCES:
- [Derived] Espiritu AI, Sy MCC, Anlacan VMM, Jamora RDG; Philippine CORONA Study Group Investigators. COVID-19 outcomes of 10,881 patients: retrospective study of neurological symptoms and associated manifestations (Philippine CORONA Study). J Neural Transm (Vienna). 2021 Nov;128(11):1687-1703. doi: 10.1007/s00702-021-02400-5. Epub 2021 Aug 27. PMID 34448930
- [Derived] Espiritu AI, Sy MCC, Anlacan VMM, Jamora RDG. The Philippine COVID-19 Outcomes: a Retrospective study Of Neurological manifestations and Associated symptoms (The Philippine CORONA study): a protocol study. BMJ Open. 2020 Nov 30;10(11):e040944. doi: 10.1136/bmjopen-2020-040944. PMID 33257488